CLINICAL TRIAL: NCT06009094
Title: Safety, Tolerance and Pharmacokinetics Clinical Study of VC005 in Healthy Subjects and Patients with Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YQ-M-23-02
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- VC005 Low Dose groups (Experimental)
  Interventions: Drug: VC005
- VC005 median-A Dose groups (Experimental)
  Interventions: Drug: VC005
- VC005 median-B Dose groups (Experimental)
  Interventions: Drug: VC005
- VC005 high Dose groups (Experimental)
  Interventions: Drug: VC005
- VC005 Placebo groups (Placebo Comparator)
  Interventions: Drug: VC005 Placebo

INTERVENTIONS:
Drug: VC005 — VC005 group with Local topical application
  Arms: VC005 Low Dose groups; VC005 high Dose groups; VC005 median-A Dose groups; VC005 median-B Dose groups
Drug: VC005 Placebo — VC005 Placebo group with Local topical application
  Arms: VC005 Placebo groups

SUMMARY:
This study is a single center, randomized, double-blind, Vehicle controlled,, single and multiple dose clinical study.

ELIGIBILITY:
Inclusion Criteria:

healthy subject's study:

1. Healthy male or female subjects, aged 18-45 years (including critical values);
2. Body mass index (BMI) between 18 and 26kg/m2 (including critical values), with male weight ≥ 50kg and female weight ≥ 45kg;
3. All women and men with fertility potential must be willing to use at least one efficient method of contraception from the signing of the informed consent form until 3 months after the last administration of the study drug, as detailed in Appendix 5;
4. Voluntarily participate in the experiment and sign an informed consent form;
5. Subjects who are able to communicate well with the researcher and are willing and able to comply with all planned visits, treatment plans, laboratory tests, and other research procedures

patient's study:

1. When informed consent is given, the age range is between 18 and 75 years (including the boundary value), regardless of gender;
2. Body mass index (BMI) between 18 and 26kg/m2 (including critical values), with male weight ≥ 50kg and female weight ≥ 45kg;
3. Before administration, the diagnosis of mild to moderate atopic dermatitis should be met:

   Overall Investigator Assessment (IGA) score of 2 to 3 points; Atopic dermatitis: total area of skin lesions 3% ≤ body surface area≤ 20%
4. Voluntarily sign an informed consent form (with a date), indicating that the subject has been informed of all relevant parts of the study;
5. All women and men with the possibility of childbirth must be willing to use at least one efficient method of contraception from the signing of the informed consent form until 3 months after the last administration of the study drug, as detailed in Appendix 5;
6. Subjects who are willing and able to comply with planned visits and treatment plans, laboratory tests, and other research procedures

Exclusion Criteria:

healthy subject's study:

1. Suspected of being allergic to the study drug or any component of the study drug, or having an allergic constitution;
2. Those who have received the vaccine within 2 weeks before administration or plan to receive the vaccine during the study period;
3. Screening for individuals who have undergone any surgery within the previous 6 months;
4. Those who participated in blood donation within the first 3 months of screening and had a blood donation volume of ≥ 400 mL, or received blood transfusion (excluding female physiological blood loss);
5. Female subjects of childbearing age had unprotected sexual intercourse with their opposite sex partner within 14 days prior to screening;
6. Screening of clinical trial participants (including excipient groups) who have participated in any drug or medical device within the first 3 months;
7. Pregnant and lactating women;
8. Patients with difficulty in blood collection or inability to tolerate venous puncture, and those with a history of needle and blood fainting;
9. Those who smoke ≥ 5 cigarettes per day within the first 3 months of screening, and cannot stop using any tobacco products from the end of screening to enrollment and during the trial period;
10. Those who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) within the first 3 months of screening, or who cannot abstain from alcohol during the trial period;
11. Other situations where the researcher determines that it is not suitable to participate in the experiment.

patient's study:

1. Suspected of being allergic to the study drug or any component of the study drug, or having an allergic constitution;
2. Those who have received the vaccine within 2 weeks before administration or plan to receive the vaccine during the study period;
3. Screening for individuals who have undergone any surgery within the previous 6 months;
4. Those who participated in blood donation within the first 3 months of screening and had a blood donation volume of ≥ 400 mL, or received blood transfusion (excluding female physiological blood loss);
5. Screening of clinical trial participants (including excipient groups) who have participated in any drug or medical device within the first 3 months;
6. Pregnant and lactating women;
7. Patients with difficulty in blood collection or inability to tolerate venous puncture, and those with a history of needle and blood fainting;
8. Those who smoke ≥ 5 cigarettes per day within the first 3 months of screening, and cannot stop using any tobacco products from the end of screening to enrollment and during the trial period;
9. Those who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) within the first 3 months of screening, or who cannot abstain from alcohol during the trial period;
10. Other situations where the researcher determines that it is not suitable to participate in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax） | Day2,Day 4,Day17,Day31

SECONDARY OUTCOMES:
Changes in EASI（Eczema area and severity index） from baseline | Week 2,Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Chinese Academy of Medical Sciences Hospital of Skin Disease
Locations (1):
- Chinese Academy of Medical Sciences Hospital of Skin Disease, Nanjing, Jiangsu, China